CLINICAL TRIAL: NCT00646555
Title: Evaluation of Angiogenesis Parameters and Tumor Markers in Inflammatory Breast Cancer Specimens
Brief Title: Inflammatory Breast Cancer, Tumor Markers, and Factors Associated With Angiogenesis
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904051; 04-C-N051; NCT00073567 (obsolete NCT alias); NCT00899314 (obsolete NCT alias)
Record Dates: First submitted 2008-03-27; First posted 2008-03-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-10

CONDITIONS: Breast Neoplasms
Keywords: Tissue Samples; VEGF Receptors; VEGF; Microvessel Density; Hypoxia Inducible Factor; Inflammatory Breast Cancer; IBC
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms

SUMMARY:
This study, conducted by the NCI and the George Washington University Medical Center (GWUMC), will examine breast tissue from patients with inflammatory breast cancer (IBC) for tumor markers and factors associated with angiogenesis. Angiogenesis is the formation of new blood vessels that is essential for tumor growth and spread. IBC is an extremely rare, aggressive form of breast cancer that disproportionately affects young women. The risk factors for IBC, its cause, and how it develops are unknown, but the disease appears to involve a high degree of angiogenesis.

Tissue specimens for this study will be obtained from GWUMC's Inflammatory Breast Cancer Registry and Biospecimen Repository. The registry was established to develop a national registry of patients with IBC that includes standardized clinical, epidemiological, and pathological information, along with disease recurrence and survival data.

For this study, tissue specimens from the repository will be tested for biological markers and angiogenesis parameters to help in the classification of the tumors. Biological markers (such as estrogen receptor, progesterone receptor, the p53 gene, and others) and angiogenesis parameters (such as various proteins involved in vessel formation) will be examined to determine their prevalence in tissue specimens and their relationship to patient survival. When possible, the findings will be compared with non-IBC tissue samples.

DETAILED DESCRIPTION:
Inflammatory breast carcinoma (IBC) is an extremely rare, aggressive form of breast cancer that disproportionately affects young women. The risk factors and pathogenesis of these tumors are unknown and it is unclear whether tumors showing various clinical, pathological or molecular features behave differently. IBC appears to be a highly angiogenic tumor. In this study, tumor markers and parameters of angiogenesis will be further investigated in IBC.

The Inflammatory Breast Cancer Registry and Biospecimen Repository is a project funded by a grant from the Department of Defense to Paul H. Levine at GWUMC. The purpose of the registry is to develop a national registry of patients with IBC that will contain standardized clinical, epidemiological, and pathological information, along with recurrence and survival data. The goal is to obtain specimens from approximately 150 patients with IBC. The data in the registry and repository will be made available to researchers to aid in the development of a clinicopathological diagnosis of IBC. Investigators at GWUMC will consent recruited patients and collect clinical data. Subjects will not be recruited, evaluated, or monitored at the NCI. The GWUMC IRB will oversee human subjects protection issues. All samples obtained from GWUMC will be blinded and coded to the NCI investigators. In addition to the samples from George Washington University, we will obtain 150 control samples from the National Cancer Institute Cooperative Breast Cancer Tissue Resource. These samples were not available when this protocol was first submitted.

In collaboration with George Washington University Medical Center (GWUMC), we plan to test tissue specimens collected in the IBC registry and biospecimen repository. We will obtain frozen tissue (tissue and/or normal) and paraffin-embedded tissue blocks from each case. Genetic testing will not be performed on any of the samples. One pathologist reviews cases for grade and lymphovascular invasion (LVI) based on H& E staining. Specimens will be tested for biological markers associated with IBC to help in classification of these tumors. These include ER, E-cadherin, podoplanin, ReIB, RhoC and vasodilator-stimulated phosphoprotein (VASP). Angiogenesis parameters will also be evaluated. These include hypoxia-inducible factor 1 alpha (HIF-1 alpha), vascular endothelial growth factor D (VEGF-D) protein expression, VEGF-C protein expression, VEGF-receptor 2 (VEGFR-2, Kdr) or VEGF-receptor 3 (VEGFR-3, flt-4).

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with inflammatory breast cancer.

Age greater than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2003-11-20; Study Completion 2012-04-10

CONTACTS AND LOCATIONS:
Overall Officials: Amy Subar, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- GW University Medical Center GW Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Folkman J. Angiogenesis and apoptosis. Semin Cancer Biol. 2003 Apr;13(2):159-67. doi: 10.1016/s1044-579x(02)00133-5. PMID 12654259
- [Background] Weidner N, Semple JP, Welch WR, Folkman J. Tumor angiogenesis and metastasis--correlation in invasive breast carcinoma. N Engl J Med. 1991 Jan 3;324(1):1-8. doi: 10.1056/NEJM199101033240101. PMID 1701519
- [Background] Gasparini G, Weidner N, Bevilacqua P, Maluta S, Dalla Palma P, Caffo O, Barbareschi M, Boracchi P, Marubini E, Pozza F. Tumor microvessel density, p53 expression, tumor size, and peritumoral lymphatic vessel invasion are relevant prognostic markers in node-negative breast carcinoma. J Clin Oncol. 1994 Mar;12(3):454-66. doi: 10.1200/JCO.1994.12.3.454. PMID 7509851